CLINICAL TRIAL: NCT05022290
Title: Comparison of Double-syringe vs Single-syringe Technique of Adenosine Administration for Termination of Regular-narrow Complex Tachycardia: A Randomized, Controlled Trial
Brief Title: Double-syringe vs Single-syringe Technique of Adenosine for Termination of Regular Narrow Complex Tachycardia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Praew Kotruchin, Associate professor, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HE631158
Record Dates: First submitted 2021-08-21; First posted 2021-08-26 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Supraventricular Tachycardia
Keywords: adenosine; tachycardia; single bolus; emergency; Asian
MeSH Terms: conditions — Tachycardia, Supraventricular; Tachycardia; Emergencies

STUDY DESIGN:
Intervention Model Description: In a randomized controlled trial, participants will be allocated into 2 groups. Each group receives adenosine with the same dosage but different methods of administration.
Who Masked: Participant
Masking Description: There will be an opaque fabric shade that covered the participant's right upper arm during treatment that does not allow them to see the methods of drug administration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single-syringe technique (Experimental): Patients in this arm will receive adenosine in a single syringe, diluted with normal saline up to 20 ml. The dosage of adenosine is according to the recommendation of ACLS guidelines, which recommended 6 mg as the first dose and 12 mg as the subsequent dose if SVT can not be terminated by the first dose.
  Interventions: Procedure: Single-syringe diluted with normal saline technique
- Double-synring technique (Active Comparator): Patients in this arm will receive adenosine using a double syringe, the first syringe contains only adenosine and the second syringe contains only normal saline 20 ml. Both syringes are connected to each other, and to the patient's IV portal with a stopcock. The administration must be done by two nurses one after another, adenosine syringe is injected first, then follow by normal saline. The dosage of adenosine is according to the recommendation of ACLS guidelines, which recommended 6 mg as the first dose and 12 mg as the subsequent dose if SVT can not be terminated by the first dose.
  Interventions: Procedure: Single-syringe diluted with normal saline technique

INTERVENTIONS:
Procedure: Single-syringe diluted with normal saline technique — Adenosine is mixed with normal saline up to 20 ml in a single syringe before administering to the patient by the IV bolus method.

SUMMARY:
Adenosine has been discovered since 1929 and used in the acute treatment of arrhythmias. It uses as a therapeutic diagnosis in patients with regular narrow QRS complex tachyarrhythmias. The conventional method of adenosine administration is the double syringe technique (DST). However, it consumes a lot of resources including two syringes, a stopcock, an extension tube, and needs 2 nurses to administer. An observational study found that a single syringe technique (adenosine diluted with normal saline up to 20 ml) was as effective as a double syringe technique. However, there is no randomized control trial for proving its efficacy.

DETAILED DESCRIPTION:
Supraventricular tachycardia (SVT) is the most common tachyarrhythmias in young adults, children, and infants. The most common type in adults is the atrioventricular nodal reentrant tachycardia (AVNRT) and the incidence is 35 per 10,000 person-years or 2.29 per 1000 persons.

The treatment approach of SVT is based on hemodynamical stability. The synchronized cardioversion is recommended for hemodynamically unstable patients, on the other hand, the vagal maneuvers and medications are considered for patients with stable hemodynamic.

To date, the 2019 ESC guideline for the management of supraventricular tachycardia stated that adenosine is still the first medication for acute therapy in patients with SVT if the vagal maneuver fails or is contraindicated. A systematic review in 2021 showed that adenosine is equally efficacious for treating SVT, but it is safer than intravenous calcium channel blockers due to a shorter half-life.

Few studies reported that the effectiveness of conventional vagal maneuvers, namely, carotid sinus massage in SVT termination was around 19 to 54% when properly done. The enhanced method of vagal maneuver or named the modified syringe technique was performed by blowing into a 10 mL syringe to move the plunger, the success conversion rate of SVT was a little better than the convention technique (43% vs 17%). Therefore, adenosine is still crucial in the acute therapy of SVT in an emergency setting.

Adenosine has been discovered since 1929 and used in the acute treatment of arrhythmias. It was used as a therapeutic diagnosis in patients with regular narrow QRS complex tachyarrhythmias and it is also helpful in treating some type of regular wide QRS complex tachyarrhythmias (differentiate between SVT with aberrancy/bundle branch block and ventricular tachycardia).

Adenosine, an endogenous purine nucleoside, is the first drug of choice to terminate SVT. The pharmacological response of adenosine is mediated through cardiac adenosine type 1 (A1) receptors and has a dose-response relationship. It prolongs atrioventricular (AV) conduction and results in transient AV block that is responsible for tachyarrhythmia termination. The dosages for the peripheral intravascular (IV) route are 6 mg and follow by 12 mg if the first dose is failed.2 To achieve rhythm conversion, the injection should be performed as a rapid bolus with immediate saline flush through large veins (e.g. antecubital) in 1-2 seconds, because adenosine is rapidly metabolized by enzymatic deamination to inactive inosine within seconds, and achieve end-organ effects within 20-30 seconds.2 This conventional method of adenosine administration is well-known as the double syringe technique (DST). The repeat dose is safe when administered at least 1 minute after the first dose. The success rate of adenosine in terminating SVT was greater than 90% approximately.

The potential side effects of adenosine are transient AV block, flushing, chest pain, or dyspnea, AF can be initiated or worsened in case of preexcitation existing, premature ventricular tachycardias (PVCs)/ventricular tachycardia (VT), bronchospasm (rare), or coronary steal.5 In addition, Adenosine should be excluded or used with caution in patients with these conditions (e.g. AV block greater than first degree or sinoatrial (SA) node dysfunction, reactive airway disease, concomitant use of verapamil or digoxin, and Wolff-Parkinson-White (WPW) syndrome).5

The DST requires a two-way stopcock which may not stock in some workplaces e.g. emergency medical services (EMS) and need the nursing staff to coordinate their actions administering the drug and flush simultaneously. In the real world, small hospitals had a transient shortage of medical equipment supply e.g. syringes. The convenient method which combined adenosine and 15 mL of normal saline in one syringe was firstly proposed in the non-blind, randomized prospective study between 1999 to 2001 and published the full original article in the Korean language since 2003 by Choi SC et al. This trial demonstrated the success rate of the convenient method was higher than the standard method (85.7 vs 80%), but it's not statistically significant, in addition, the average of total administering doses, and the complication of the convenient and standard method was not statistically different.

Nearly two decades later, Marc McDowell et al. conducted a single-center, prospective, observational study with setting a 20% non-inferiority margin demonstrated that the successful conversion of SVT in the first dose (73.1 vs 40.7%) and up to three doses (100 vs 70.4%) in the single syringe technique (SST) and DST respectively. And they didn't found any serious adverse effects e.g. dyspnea, bradycardia, or asystole. Unfortunately, superiority testing was not performed due to the limiting sample size.

Therefore, we hypothesized that the SST is non-inferior to the DST for terminating stable SVT, by comparison, a rate of successful conversion of SVT at the first 6 mg-dose of adenosine and the total average dosage of adenosine administered. And we also aimed to compare the rate of side effects between both techniques of intravenous adenosine in those diagnosed with stable SVT.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-80 years old
* EKG shows regular rhythm, narrow QRS complex tachyarrhythmias (QRS complex <0.12 msec, and rate >150 beats per minute; bpm)
* Pulse can be palpated
* The tachycardia is not terminated by a vagal maneuver.

Exclusion Criteria:

* Acute asthmatic attack
* Pregnant or tendency to be pregnant
* Acute heart failure
* Acute chest pain
* Alteration of consciousness
* Hypotension
* Presenting of signs of hypoperfusion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Termination of supraventricular tachycardia (SVT) | 1 minute after complete administration of adenosine intravenously
  The outcome is achieved when doctor in charge determine that the supraventricular tachycardia is terminated by administration of adenosine with the EKG after treatment showing sinus rhythm.

SECONDARY OUTCOMES:
Total dose of adenosine used for termination of supraventricular tachycardia | 10 minutes after diagnosis of supraventricular tachycardia
  Calculated the total dose of adenosine administration of each patient (milligram)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Emergency medicine, Khon Kaen, Muang, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
Will decide after a complete enrollment.